CLINICAL TRIAL: NCT02297438
Title: A MULTICENTER, RANDOMIZED, DOUBLE-BLIND PHASE 3 STUDY OF PALBOCICLIB (ORAL CDK 4/6 INHIBITOR) PLUS LETROZOLE VERSUS PLACEBO PLUS LETROZOLE FOR THE TREATMENT OF PREVIOUSLY UNTREATED ASIAN POSTMENOPAUSAL WOMEN WITH ER (+), HER2 (-) ADVANCED BREAST CANCER
Brief Title: A Study Of Palbociclib (PD-0332991) + Letrozole VS. Placebo+ Letrozole For 1st Line Treatment Of Asian Postmenopausal Women With ER+/HER2- Advanced Breast Cancer [PALOMA-4]
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A5481027; NCT02297438 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Results first posted 2021-11-18 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; postmenopausal women; estrogen-receptor positive; HER2 negative; locoregionally recurrent; metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — palbociclib; Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palbociclib + Letrozole (Experimental): Palbociclib, 125mg, orally once daily on Day 1 to Day 21 of every 28-day cycle followed by 7 days off treatment in combination with Letrozole, 2.5mg, orally once daily (continuously)
  Interventions: Drug: Palbociclib; Drug: Letrozole
- Placebo + Letrozole (Active Comparator): Placebo, 125mg, orally once daily on Day 1 to Day 21 of every 28-day cycle followed by 7 days off treatment in combination with Letrozole, 2.5mg, orally once daily (continuously).
  Interventions: Drug: Placebo; Drug: Letrozole

INTERVENTIONS:
Drug: Palbociclib — Palbociclib, 125mg, orally once daily on Day 1 to Day 21 of every 28-day cycle followed by 7 days off treatment
  Other Names: PD-0332991
  Arms: Palbociclib + Letrozole
Drug: Letrozole — Letrozole, 2.5mg, orally once daily (continuously)
  Arms: Palbociclib + Letrozole
Drug: Placebo — Placebo, 125mg, orally once daily on Day 1 to Day 21 of every 28-day cycle followed by 7 days off treatment
  Arms: Placebo + Letrozole
Drug: Letrozole — Letrozole, 2.5mg, orally once daily (continuously)
  Arms: Placebo + Letrozole

SUMMARY:
The study is designed to compare the clinical benefit following treatment with letrozole in combination with Palbociclib versus letrozole in combination with placebo in Asian postmenopausal women with ER(+)/HER2(-) advanced breast cancer who have not received prior systemic anti cancer therapies for their advanced/metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult Asian women with locoregionally recurrent or metastatic disease not amenable to curative therapy
* Confirmed diagnosis of ER positive breast cancer
* No prior systemic anti-cancer therapy for advanced ER+ disease
* Postmenopausal women
* Measurable disease as per Response Evaluation Criterion in Solid Tumors [RECIST] or bone-only disease
* Eastern Cooperative Oncology Group [ECOG] 0-1
* Adequate organ and marrow function
* Patient must agree to provide tumor tissue

Exclusion Criteria:

* Confirmed diagnosis of HER2 positive disease
* Patients with advanced, symptomatic, visceral spread that are at risk of life threatening complication in the short term
* Known uncontrolled or symptomatic CNS metastases
* Prior neoadjuvant or adjuvant treatment with a non steroidal aromatase inhibitor (ie, anastrozole or letrozole) with disease recurrence while on or within 12 months of completing treatment
* Prior treatment with any CDK 4/6 inhibitor

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 340 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2025-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (53):
- China (33):
  - The First Affiliated Hospital of Bengbu Medical College/Medical Oncology Department, Bengbu, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Fujian Medical University Union Hospital/Medical Oncology Department, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Zhongshan Ophthalmic Center,Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Breast Tumor Center, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital/Oncology Department, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Provincial Tumor Hospital/Breast Internal Medicine Department, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Jilin Provincial Cancer Hospital, Changchun, Jilin
  - The First Hospital of China Medical University/Oncology Department, Shenyang, Liaoning
  - Liaoning Province Cancer Hospital, Shenyang, Liaoning
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Cancer Hospital/Breast cancer department, Tianjin, Tianjin Municipality
  - The Tumor Hospital of Yunnan Province, Kunming, Yunnan
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of College of Medicine of Zhejiang University, Center for Oncology, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing
  - 307 Hospital of PLA, Beijing
  - Beijing Cancer Hospital, Beijing
  - Peking University Third Hospital/Department of Oncology, Beijing
  - Chinese PLA General Hospital/Oncology, Beijing
  - Oncology Department, the Second Affiliated Hospital of Third Military Medical University, PLA, Chongqing
  - Fudan University Shanghai Cancer Center, Shanghai
- Hong Kong (2):
  - Department of Clinical Oncology, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Singapore (3):
  - Raffles Cancer Centre, Singapore
  - Parkway Cancer Centre, Singapore
  - Tan Tock Seng Hospital, Singapore
- Taiwan (8):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital / Internal Medicine, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Medical University Hospital/ Department of Surgery, Taipei
  - Taipei Veterans General Hospital/Surgery Department, Taipei
  - Koo Foundation, Sun Yat-Sen Cancer Center, Taipei
  - Taipei Municipal Wanfang Hospital (Managed by Taipei Medical University ), Taipei
- Thailand (7):
  - King Chulalongkorn Memorial Hospital, Pathumwan, Bangkok
  - Chula Clinical Research Center (Chula CRC), Patumwan, Bangkok
  - Department of Medicine, Faculty of Medicine, Naresuan University, Muang, Changwat Phitsanulok
  - Division of Therapeutic Radiology and Oncology, Department of Radiology, Muang, Chiang Mai
  - Ramathibodi Hospital, Mahidol University, Bangkok, Ratchathevi
  - Oncology Unit, Department of Internal Medicine, Phramongkutklao Hospital, Bangkok
  - Division of Medical Oncology, Department of Medicine,, Bangkok

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Xu B, Hu X, Li W, Sun T, Shen K, Huang C, Sriuranpong V, Ngan RK, Chia YH, Reisman A, Zhao H, Shen J, Broughton E. Patient-reported quality of life in Asian patients with ER+/HER2- advanced breast cancer treated with palbociclib plus letrozole in the PALOMA-4 trial. Chin Med J (Engl). 2024 Dec 19. doi: 10.1097/CM9.0000000000003122. Online ahead of print. PMID 39694573
- [Derived] Xu B, Hu X, Li W, Sun T, Shen K, Wang S, Cheng Y, Zhang Q, Cui S, Tong Z, Geng C, Song E, Huang CS, Sriuranpong V, Ngan RKC, Chia YH, Wang X, Zhao H. Palbociclib plus letrozole versus placebo plus letrozole in Asian postmenopausal women with oestrogen receptor-positive/human epidermal growth factor receptor 2-negative advanced breast cancer: Primary results from PALOMA-4. Eur J Cancer. 2022 Nov;175:236-245. doi: 10.1016/j.ejca.2022.08.012. Epub 2022 Sep 22. PMID 36155117
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481027&StudyName=A%20Study%20Of%20Palbociclib%20%28PD-0332991%29%20+%20Letrozole%20VS.%20Placebo+%20Letrozole%20For%201st%20Line%20Treatment%20Of%20East%20Asian%20Postmenopausal%20Women%20Wit

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a multicenter, randomized (1:1), double blind, placebo controlled, parallel group Phase 3 trial comparing the efficacy and safety of palbociclib in combination with letrozole versus placebo plus letrozole in Asian postmenopausal women with estrogen receptor positive/human epidermal growth factor receptor 2 negative advanced breast cancer.
Groups:
- Palbociclib + Letrozole: Participants were planned to receive palbociclib 125 mg orally once a day (QD) for 21 days of every 28-day cycle followed by 7 days off treatment together with letrozole 2.5 mg orally QD continuously. The maximum duration of treatment for palbociclib and for letrozole were 1872 days and 1872 days, respectively.
- Placebo + Letrozole: Participants were planned to receive placebo 125 mg orally once a day (QD) for 21 days of every 28-day cycle followed by 7 days off treatment together with letrozole 2.5 mg orally QD continuously. The maximum duration of treatment for placebo and for letrozole were 1834 days and 1834 days, respectively.
Period: Overall Study
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Started | 169 | 171
Received Treatment | 168 | 171
Completed | 0 | 0
Not Completed | 169 | 171
Not completed — Death | 79 | 86
Not completed — Lost to Follow-up | 9 | 7
Not completed — Withdrawal by Subject | 7 | 0
Not completed — Other | 9 | 5
Not completed — Ongoing | 65 | 73

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole | Total
Number analyzed (Participants) | 169 | 171 | 340
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (8.5) | 53.7 (9.1) | 53.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 171 | 340
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 169 | 171 | 340

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Based on Investigator's Assessment
Description: PFS was based on Kaplan-Meier estimates. PFS was defined as the time from the date of randomization to the date of the first documentation of objective progression of disease (PD) or death due to any cause in the absence of documented PD, whichever occurred first. PD is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) as a 20% increase in the sum of of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy), with a minimum absolute increase of 5 mm. In this outcome measure, PFS was based on investigator's assessment.
Time Frame: Randomization up to 65 months
Population: This was intent-to-treat (ITT) population, including all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 169 | 171
Months | 21.5 [16.6 to 24.9] | 13.9 [13.7 to 16.6]
Statistical Analysis 1: Comparison: Palbociclib + Letrozole vs Placebo + Letrozole; Stratified by disease site (visceral vs. non-visceral) per Randomization; Test type: Superiority; p = 0.0012, Log Rank — 1-sided p-value from the adjusted log-rank test; Hazard Ratio (HR) = 0.677, 95% CI 2-sided [0.529 to 0.867] — Assuming proportional hazards, a hazard ratio less than 1 indicates a reduction in hazard rate in favor of Palbociclib + Letrozole

2. Secondary Outcome: Progression-Free Survival (PFS) Based on Blinded Independent Central Review (BICR)
Description: PFS was based on Kaplan-Meier estimates. PFS was defined as time from the first dose of study treatment to the first documentation of objective tumor progression or to death due to any cause in the absence of documented progressive disease, whichever occurs first. In this outcome measure, PFS was based on BICR.
Time Frame: Randomization up to 65 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 169 | 171
Months | 21.6 [16.6 to 30.4] | 16.4 [13.8 to 22.2]
Statistical Analysis 1: Comparison: Palbociclib + Letrozole vs Placebo + Letrozole; Stratified by disease site (visceral versus non-visceral) per Randomization; Test type: Superiority; p = 0.14778, Log Rank — 1-sided p-value from the log-rank test; Hazard Ratio (HR) = 0.861, 95% CI 2-sided [0.651 to 1.139] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Wiht Objective Response (OR) Based on Investigator Assessment
Description: OR was defined as a complete response (CR) or partial response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 recorded from randomization until disease progression or death due to any cause. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). No new lesions. The PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No new lesions. In this outcome measure, OR was based on investigator assessment.
Time Frame: Randomization up to 65 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 169 | 171
Percentage of participants | 37.3 [30.0 to 45.0] | 31.6 [24.7 to 39.1]
Statistical Analysis 1: Comparison: Palbociclib + Letrozole vs Placebo + Letrozole; Stratified by disease site (visceral versus non-visceral) per Randomization; Test type: Superiority; p = 0.154, Fisher Exact — 1-sided p-value was from exact test; Odds Ratio (OR) = 1.301, 95% CI 2-sided [0.805 to 2.100] — An Odds Ratio >1 means better response in favor of Palbociclib + Letrozole group

4. Secondary Outcome: Percentage of Participants With Objective Response (OR) Based on Investigator Assessment (Participants With Measureable Disease at Baseline)
Description: as for outcome 3
Time Frame: Randomization up to 65 months
Population: This was intent-to-treat (ITT) population with measureable disease at baseline, including the participants, who were randomized, with measureable disease at baseline, and study drug assignment designated according to initial randomization, regardless of whether participants received study drug or received a different drug from that to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 145 | 142
Percentage of participants | 43.4 [35.2 to 51.9] | 38.0 [30.0 to 46.5]
Statistical Analysis 1: Comparison: Palbociclib + Letrozole vs Placebo + Letrozole; Stratified by disease site (visceral versus non-visceral) per Randomization; Test type: Superiority; p = 0.206, Fisher Exact — 1-sided p-value was from exact test; Odds Ratio (OR) = 1.255, 95% CI 2-sided [0.762 to 2.066] — An Odds Ratio >1 means better response in favor of Palbociclib + Letrozole group

5. Secondary Outcome: Percentage of Participants With Objective Response (OR) Based on Blinded Independent Central Review (BICR)
Description: OR was defined as a complete response (CR) or partial response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 recorded from randomization until disease progression or death due to any cause. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). No new lesions. The PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No new lesions. In this outcome measure, OR was based on BICR.
Time Frame: Randomization up to 65 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 169 | 171
Percentage of participants | 40.2 [32.8 to 48.0] | 33.9 [26.9 to 41.5]
Statistical Analysis 1: Comparison: Palbociclib + Letrozole vs Placebo + Letrozole; Stratified by disease site (visceral versus non-visceral) per Randomization; Test type: Superiority; p = 0.135, Fisher Exact — 1-sided p-value was from exact test; Odds Ratio (OR) = 1.315, 95% CI 2-sided [0.825 to 2.095] — An Odds Ratio >1 means better response in favor of Palbociclib + Letrozole group

6. Secondary Outcome: Percentage of Participants With Objective Response (OR) Based on Blinded Independent Central Review (BICR) (Participants With Measureable Disease at Baseline)
Description: as for outcome 5
Time Frame: Randomization up to 65 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 128 | 131
Percentage of participants | 52.3 [43.3 to 61.2] | 43.5 [34.9 to 52.4]
Statistical Analysis 1: Comparison: Palbociclib + Letrozole vs Placebo + Letrozole; Stratified by disease site (visceral versus non-visceral) per Randomization; Test type: Superiority; p = 0.117, Fisher Exact — 1-sided p-value was from exact test; Odds Ratio (OR) = 1.392, 95% CI 2-sided [0.825 to 2.346] — An Odds Ratio >1 means better response in favor of Palbociclib + Letrozole group

7. Secondary Outcome: Duration of Response (DOR) Based on Investigator Assessment (Participants With Objective Disease Response)
Description: DOR was defined as the time from the first documentation of objective tumor response (complete response [CR] or partial response [PR]) to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first. DOR data was censored on the date of the last tumor assessment on study for participants who did not have objective tumor progression and who did not die due to any cause while on study. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). No new lesions. The PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No new lesions. In this outcome measure, DOR was based on investigator assessment.
Time Frame: Randomization up to 65 months
Population: This was intent-to-treat (ITT) population with objective disease response, including all participants who were randomized, with objective disease response and study drug assignment designated according to initial randomization, regardless of whether participants received study drug or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 63 | 54
Months | 22.4 [19.4 to 56.2] | 19.4 [13.8 to 24.4]

8. Secondary Outcome: Duration of Response (DOR) Based on Blinded Independent Central Review (BICR) (Participants With Objective Disease Response)
Description: DOR was defined as the time from the first documentation of objective tumor response (complete response [CR] or partial response [PR]) to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first. DOR data was censored on the date of the last tumor assessment on study for participants who did not have objective tumor progression and who did not die due to any cause while on study. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). No new lesions. The PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No new lesions. In this outcome measure, DOR was based on BICR.
Time Frame: Randomization up to 65 months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 68 | 58
Months | 30.3 [19.4 to NA] — As 50% participants in this analysis set was censored, the upper bound of 95% confidence interval was not reached. | 24.9 [11.5 to 36.1]

9. Secondary Outcome: Percentage of Participants With Disease Control/Clinical Benefit Response (DC/CBR) Based on Investigator Assessment
Description: DC/CBR was defined as CR, PR, or stable disease (SD) >=24 weeks according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1) recorded in the time period between randomization and disease progression or death to any cause. CR was defined as complete disappearance of all target lesions except for nodal disease. All target nodes must decrease to normal size (short axis <10 mm). No new lesions. The PR was defined as >=30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No new lesions. SD was defined as not qualifying for CR, PR, PD. PD is defined using RECIST v1.1 as a 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed, with a minimum absolute increase of 5 mm. In this outcome measure, DC/CBR was based on investigator assessment.
Time Frame: Randomization up to 65 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 169 | 171
Percentage of participants | 79.3 [72.4 to 85.1] | 80.1 [73.3 to 85.8]
Statistical Analysis 1: Comparison: Palbociclib + Letrozole vs Placebo + Letrozole; Stratified by disease site (visceral versus non-visceral) per Randomization; Test type: Superiority; p = 0.471, Fisher Exact — 1-sided p-value was from exact test; Odds Ratio (OR) = 0.945, 95% CI 2-sided [0.533 to 1.673] — An Odds Ratio >1 means better response in favor of Palbociclib + Letrozole group

10. Secondary Outcome: Percentage of Participants With Disease Control/Clinical Benefit Response (DC/CBR) Based on Investigator Assessment (Participants With Measureable Disease at Baseline)
Description: DC/CBR was defined as CR, PR, or stable disease (SD) >=24 weeks according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1) recorded in the time period between randomization and disease progression or death to any cause. CR was defined as complete disappearance of all target lesions except for nodal disease. All target nodes must decrease to normal size (short axis <10 mm). No new lesions. The PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No new lesions. SD was defined as not qualifying for CR, PR, PD. PD is defined using RECIST v1.1 as a 20% increase in the sum of of diameters of target measurable lesions above the smallest sum observed, with a minimum absolute increase of 5 mm. In this outcome measure, DC/CBR was based on investigator assessment.
Time Frame: Randomization up to 65 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 145 | 142
Percentage of participants | 77.9 [70.3 to 84.4] | 79.6 [72.0 to 85.9]
Statistical Analysis 1: Comparison: Palbociclib + Letrozole vs Placebo + Letrozole; Stratified by disease site (visceral versus non-visceral) per Randomization; Test type: Superiority; p = 0.383, Fisher Exact — 1-sided p-value was from exact test; Odds Ratio (OR) = 0.878, 95% CI 2-sided [0.474 to 1.621] — An Odds Ratio >1 means better response in favor of Palbociclib + Letrozole group

11. Secondary Outcome: Percentage of Participants With Disease Control/Clinical Benefit Response (DC/CBR) Based on Blinded Independent Central Review (BICR)
Description: DC/CBR was defined as CR, PR, or stable disease (SD) >=24 weeks according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1) recorded in the time period between randomization and disease progression or death to any cause. CR was defined as complete disappearance of all target lesions except for nodal disease. All target nodes must decrease to normal size (short axis <10 mm). No new lesions. The PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No new lesions. SD was defined as not qualifying for CR, PR, PD. PD is defined using RECIST v1.1 as a 20% increase in the sum of of diameters of target measurable lesions above the smallest sum observed, with a minimum absolute increase of 5 mm. In this outcome measure, DC/CBR was based on BICR.
Time Frame: Randomization up to 65 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 169 | 171
Percentage of participants | 76.9 [69.8 to 83.0] | 73.1 [65.8 to 79.6]
Statistical Analysis 1: Comparison: Palbociclib + Letrozole vs Placebo + Letrozole; Stratified by disease site (visceral versus non-visceral) per Randomization; Test type: Superiority; p = 0.248, Fisher Exact — 1-sided p-value was from exact test; Odds Ratio (OR) = 1.227, 95% CI 2-sided [0.725 to 2.082] — An Odds Ratio >1 means better response in favor of Palbociclib + Letrozole group

12. Secondary Outcome: Percentage of Participants With Disease Control/Clinical Benefit Response (DC/CBR) Based on Blinded Independent Central Review (BICR) (Participants With Measureable Disease at Baseline)
Description: as for outcome 11
Time Frame: Randomization up to 65 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 128 | 131
Percentage of participants | 78.1 [70.0 to 84.9] | 71.8 [63.2 to 79.3]
Statistical Analysis 1: Comparison: Palbociclib + Letrozole vs Placebo + Letrozole; Stratified by disease site (visceral versus non-visceral) per Randomization; Test type: Superiority; p = 0.189, Fisher Exact — 1-sided p-value was from exact test; Odds Ratio (OR) = 1.349, 95% CI 2-sided [0.731 to 2.509] — An Odds Ratio >1 means better response in favor of Palbociclib + Letrozole group

13. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of randomization to date of death due to any cause. In the absence of confirmation of death, survival time was censored to last date the participant was known to be alive. OS was assessed using Kaplan-Meier methods.
Time Frame: Randomization up to 65 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 169 | 171
Months | 51.7 [43.0 to NA] — As 50% participants in this analysis set was censored, the upper bound of 95% confidence interval was not reached. | 51.5 [41.0 to NA] — As 50% participants in this analysis set was censored, the upper bound of 95% confidence interval was not reached.
Statistical Analysis 1: Comparison: Palbociclib + Letrozole vs Placebo + Letrozole; Stratified by disease site (visceral versus non-visceral) per Randomization; Test type: Superiority; p = 0.36502, Log Rank — 1-sided p-value was from exact test; Hazard Ratio (HR) = 0.947, 95% CI 2-sided [0.698 to 1.286] — Assuming Cox proportional hazards, hazard ratio less than 1 indicates reduction in hazard rate in favor of Palbociclib + Letrozole

14. Secondary Outcome: 1-Year, 2-Year and 3-Year Survival Probability
Description: OS was defined as the time from date of randomization to date of death due to any cause. In the absence of confirmation of death, survival time was censored to last date the participant was known to be alive. The 1-year survival probability was estimated using the Kaplan-Meier method and a 2-sided 95% confidence interval (CI) for the log [-log(1 year survival probability)] was be calculated using a normal approximation, and then back transformed to give a CI for the 1-year survival probability itself. The 2-year, and 3-year survival probabilities were estimated similarly.
Time Frame: Randomization up to 65 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 169 | 171
Percentage of participants
  1-year survival probability | 92.8 [87.6 to 95.8] | 90.5 [85.0 to 94.1]
  2-year survival probability | 80.3 [73.3 to 85.6] | 78.0 [71.0 to 83.6]
  3-year survival probability | 67.1 [59.1 to 73.8] | 60.6 [52.7 to 67.5]

15. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (All Causalities)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious AE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Participants were counted only once per treatment in each row.
Time Frame: Randomization up to 65 months
Population: This was as-treated (AT) population, including all participants who received at least 1 dose of study medication, with treatment assignments designated according to actual study treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 168 | 171
Participants
  Participants with AEs | 168 | 155
  Participants with SAEs | 26 | 16
  Participants with Grade 3 or 4 AEs | 152 | 38
  Participants with Grade 5 AEs | 4 | 2
  Participants discontinued study due to AEs | 13 | 5
  Participants discontinued Palbociclib/Placebo or Letrozole due to AEs | 11 | 4
  Participants discontinued Palbociclib/Placebo due to AEs | 11 | 4
  Participants discontinued Letrozole due to AEs | 10 | 3
  Participants temporarily discontinued Palbociclib/Placebo due to AEs | 136 | 17
  Participants temporarily discontinued Letrozole due to AEs | 11 | 9
  Participants with dose reduction of Palbociclib/Placebo due to AEs | 16 | 2
  Participants with dose reduction and temporary discontinuations of Palbociclib/Placebo due to AEs | 38 | 2

16. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (Treatment Related)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious AE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to treatment was assessed by the investigator (Yes/No). Participants were counted only once per treatment in each row.
Time Frame: Randomization up to 65 months
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 168 | 171
Participants
  Participants with AEs | 167 | 123
  Participants with SAEs | 8 | 3
  Participants with Grade 3 or 4 AEs | 149 | 18
  Participants with Grade 5 AEs | 1 | 0
  Participants discontinued study due to AEs | 6 | 2
  Participants discontinued Palbociclib/Placebo or Letrozole due to AEs | 5 | 2
  Participants discontinued due to AEs related to Palbociclib/Placebo | 5 | 2
  Participants discontinued due to AEs related to Letrozole | 1 | 0
  Participants temporarily discontinued Palbociclib/Placebo due to AEs | 132 | 11
  Participants temporarily discontinued Letrozole due to AEs | 7 | 5
  Participants with dose reduction of Palbociclib/Placebo due to AEs | 15 | 2
  Participants with dose reduction and temporary discontinuations of Palbociclib/Placebo due to AEs | 37 | 2

17. Secondary Outcome: Number of Participants With Postbaseline Laboratory Abnormalities of Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 or 4 (Participants With Baseline Laboratory Abnormalities of CTCAE Grade <=2) - Hematology
Description: The laboratory results were graded according to the National Cancer Institute (NCI) CTCAE v4.0 severity grade. Shift tables were provided to examine the distribution of laboratory toxicities. The following hematology parameters had met the criteria of CTCAE grade shift change from Grade <=2 at baseline to Grade 3 or 4 post baseline: neutrophils (absolute), white blood cells, platelets, anemia and hemoglobin increased.
Time Frame: Randomization up to 65 months
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 168 | 171
Participants
  Neutrophils (absolute) | 143 | 2
  White blood cells | 77 | 1
  Platelets | 13 | 1
  Anemia | 10 | 3
  Hemoglobin increased | 3 | 0

18. Secondary Outcome: Number of Participants With Postbaseline Laboratory Abnormalities of Common Terminology Criteria for Adverse Events(CTCAE) Grade 3 or 4 (Participants With Baseline Laboratory Abnormalities of CTCAE Grade <=2) - Chemistry
Description: The laboratory results were graded according to the National Cancer Institute (NCI) CTCAE v4.0 severity grade. Shift tables were provided to examine the distribution of laboratory toxicities. The following chemistry parameters had met the criteria of CTCAE grade shift change from Grade <=2 at baseline to Grade 3 or 4 post baseline: alanine aminotransferase (ALT), alkaline phosphatase, aspartate aminotransferase (AST), bilirubin (total), creatinine, hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, and hyponatremia.
Time Frame: Randomization up to 65 months
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 168 | 171
Participants
  ALT | 9 | 1
  Alkaline phosphatase | 0 | 2
  AST | 9 | 6
  Bilirubin (total) | 2 | 2
  Creatinine | 1 | 0
  Hypercalcemia | 1 | 2
  Hyperglycemia: number analyzed (Participants) | 167 | 171
  Hyperglycemia | 1 | 1
  Hyperkalemia | 1 | 0
  Hypermagnesemia | 10 | 8
  Hypernatremia | 2 | 1
  Hypoalbuminemia | 0 | 0
  Hypocalcemia | 1 | 1
  Hypoglycemia: number analyzed (Participants) | 167 | 171
  Hypoglycemia | 0 | 1
  Hypokalemia | 3 | 6
  Hypomagnesemia | 3 | 1
  Hyponatremia | 11 | 2

19. Secondary Outcome: Trough Plasma Concentration of Palbociclib
Description: Summary of palbociclib trough concentrations
Time Frame: Pre-dose on Day 14 of Cycle 1 and Cycle 2
Population: This was a subset of as-treated (AT) population (participants who received at least 1 dose of study medication, with treatment assignments designated according to actual study treatment received), including all participants who are treated with palbociclib and have at least 1 measured plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Palbociclib + Letrozole
Number analyzed (Participants) | 143
ng/mL
  Cycle 1: number analyzed (Participants) | 128
  Cycle 1 | 81.1 (29)
  Cycle 2: number analyzed (Participants) | 114
  Cycle 2 | 77.4 (43)
  Average trough concentration | 80.2 (36)

20. Secondary Outcome: Model Estimated Mean Change From Baseline in Euro Quality of Life 5-Dimension Scale (EQ-5D) Index Scores
Description: The EQ-5D is a 6-item instrument designed to assess health status in terms of a single index value or utility score. It consists of 5 descriptors of current health state (mobility, self care, usual activities, pain/discomfort, and anxiety/depression); a participant was asked to rate each state on a 3 level scale (1=no problem, 2=some problem, and 3=extreme problem) with higher levels indicating greater severity/impairment.
Time Frame: Baseline up to Cycle 65 Day 1
Population: This was a subset of intent-to-treat (ITT) population (participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or received a different drug from that to which they were randomized), who had both baseline and who completed all 5 items needed to calculated the index-based summary score ata the respective cycle.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 166 | 171
Units on a scale
  Cycle 2 Day 1 | 0.013 [-0.01 to 0.03] | 0.014 [-0.01 to 0.03]
  Cycle 3 Day 1 | 0.012 [-0.01 to 0.03] | 0.011 [-0.01 to 0.03]
  Cycle 5 Day 1 | 0.010 [-0.01 to 0.03] | 0.005 [-0.01 to 0.03]
  Cycle 7 Day 1 | 0.008 [-0.01 to 0.03] | 0.000 [-0.02 to 0.02]
  Cycle 9 Day 1 | 0.006 [-0.02 to 0.03] | -0.006 [-0.03 to 0.02]
  Cycle 11 Day 1 | 0.004 [-0.02 to 0.03] | -0.012 [-0.04 to 0.01]
  Cycle 13 Day 1 | 0.02 [-0.02 to 0.03] | -0.017 [-0.04 to 0.01]
  Cycle 15 Day 1 | 0.000 [-0.03 to 0.03] | -0.023 [-0.05 to 0.01]
  Cycle 17 Day 1 | -0.002 [-0.03 to 0.03] | -0.029 [-0.06 to 0.00]
  Cycle 19 Day 1 | -0.004 [-0.04 to 0.03] | -0.034 [-0.07 to 0.00]
  Cycle 21 Day 1 | -0.006 [-0.04 to 0.03] | -0.040 [-0.08 to 0.00]
  Cycle 23 Day 1 | -0.008 [-0.05 to 0.03] | -0.045 [-0.08 to -0.01]
  Cycle 25 Day 1 | -0.010 [-0.05 to 0.03] | -0.051 [-0.09 to -0.01]
  Cycle 27 Day 1 | -0.012 [-0.05 to 0.03] | -0.057 [-0.10 to -0.01]
  Cycle 29 Day 1 | -0.014 [-0.06 to 0.03] | -0.062 [-0.11 to -0.02]
  Cycle 31 Day 1 | -0.016 [-0.06 to 0.03] | -0.068 [-0.12 to -0.02]
  Cycle 33 Day 1 | -0.018 [-0.07 to 0.03] | -0.074 [-0.13 to -0.02]
  Cycle 35 Day 1 | -0.020 [-0.07 to 0.03] | -0.079 [-0.13 to -0.02]
  Cycle 37 Day 1 | -0.022 [-0.08 to 0.03] | -0.085 [-0.14 to -0.03]
  Cycle 39 Day 1 | -0.024 [-0.08 to 0.03] | -0.090 [-0.15 to -0.03]
  Cycle 41 Day 1 | -0.027 [-0.09 to 0.03] | -0.096 [-0.16 to -0.03]
  Cycle 43 Day 1 | -0.029 [-0.09 to 0.04] | -0.102 [-0.17 to -0.03]
  Cycle 45 Day 1 | -0.031 [-0.10 to 0.04] | -0.107 [-0.18 to -0.04]
  Cycle 47 Day 1 | -0.033 [-0.10 to 0.04] | -0.113 [-0.19 to -0.04]
  Cycle 49 Day 1 | -0.035 [-0.11 to 0.04] | -0.119 [-0.20 to -0.04]
  Cycle 51 Day 1 | -0.037 [-0.11 to 0.04] | -0.124 [-0.20 to -0.04]
  Cycle 53 Day 1 | -0.039 [-0.12 to 0.04] | -0.130 [-0.21 to -0.05]
  Cycle 55 Day 1 | -0.041 [-0.12 to 0.04] | -0.136 [-0.22 to -0.05]
  Cycle 57 Day 1 | -0.043 [-0.13 to 0.04] | -0.141 [-0.23 to -0.05]
  Cycle 59 Day 1 | -0.045 [-0.13 to 0.04] | -0.147 [-0.24 to -0.05]
  Cycle 61 Day 1 | -0.047 [-0.14 to 0.04] | -0.152 [-0.25 to -0.06]
  Cycle 63 Day 1 | -0.049 [-0.14 to 0.04] | -0.158 [-0.26 to -0.06]
  Cycle 65 Day 1 | -0.051 [-0.15 to 0.04] | -0.164 [-0.27 to -0.06]
Statistical Analysis 1: Comparison: Palbociclib + Letrozole vs Placebo + Letrozole; The analysis based on repeated measures mixed-effects model with an intercept term, treatment, time, treatment-by-time, and baseline as covariate; Test type: Superiority; p = 0.1914, Mixed effects model; Mean = 0.031, 95% CI 2-sided [-0.02 to 0.08] — A positive change indicates improvement from baseline and a negative change indicates deterioration

21. Secondary Outcome: Model Estimated Mean Change From Baseline in Euro Quality of Life (EQ) Visual Analog Scale (VAS) Scores
Description: The EQ VAS recorded the participant's self rated questionnaire to assess generic health status on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state). Published weights were available that allow for the creation of a single summary score.
Time Frame: Baseline up to Cycle 65 Day 1
Population: as for outcome 20
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 166 | 171
Units on a scale
  Cycle 2 Day 1 | 3.047 [1.53 to 4.57] | 1.861 [0.35 to 3.37]
  Cycle 3 Day 1 | 3.125 [1.62 to 4.63] | 1.815 [0.32 to 3.31]
  Cycle 5 Day 1 | 3.279 [1.79 to 4.77] | 1.724 [0.24 to 3.21]
  Cycle 7 Day 1 | 3.434 [1.94 to 4.92] | 1.634 [0.16 to 3.11]
  Cycle 9 Day 1 | 3.589 [2.09 to 5.09] | 1.543 [0.05 to 3.03]
  Cycle 11 Day 1 | 3.743 [2.22 to 5.26] | 1.452 [-0.06 to 2.97]
  Cycle 13 Day 1 | 3.898 [2.35 to 5.45] | 1.361 [-0.19 to 2.92]
  Cycle 15 Day 1 | 4.052 [2.46 to 5.65] | 1.271 [-0.34 to 2.88]
  Cycle 17 Day 1 | 4.207 [2.56 to 5.85] | 1.180 [-0.49 to 2.85]
  Cycle 19 Day 1 | 4.362 [2.65 to 6.07] | 1.089 [-0.65 to 2.83]
  Cycle 21 Day 1 | 4.516 [2.74 to 6.29] | 0.998 [-0.83 to 2.82]
  Cycle 23 Day 1 | 4.671 [2.82 to 6.52] | 0.908 [-1.01 to 2.82]
  Cycle 25 Day 1 | 4.826 [2.89 to 6.76] | 0.817 [-1.20 to 2.83]
  Cycle 27 Day 1 | 4.980 [2.96 to 7.00] | 0.726 [-1.39 to 2.84]
  Cycle 29 Day 1 | 5.135 [3.02 to 7.25] | 0.635 [-1.59 to 2.86]
  Cycle 31 Day 1 | 5.289 [3.08 to 7.50] | 0.545 [-1.79 to 2.88]
  Cycle 33 Day 1 | 5.444 [3.13 to 7.76] | 0.454 [-1.99 to 2.90]
  Cycle 35 Day 1 | 5.599 [3.18 to 8.02] | 0.363 [-2.20 to 2.93]
  Cycle 37 Day 1 | 5.753 [3.23 to 8.28] | 0.272 [-2.42 to 2.96]
  Cycle 39 Day 1 | 5.908 [3.28 to 8.54] | 0.182 [-2.63 to 2.99]
  Cycle 41 Day 1 | 6.063 [3.32 to 8.81] | 0.091 [-2.85 to 3.03]
  Cycle 43 Day 1 | 6.217 [3.36 to 9.07] | 0.000 [-3.06 to 3.06]
  Cycle 45 Day 1 | 6.372 [3.40 to 9.34] | -0.091 [-3.28 to 3.10]
  Cycle 47 Day 1 | 6.526 [3.44 to 9.61] | -0.181 [-3.51 to 3.14]
  Cycle 49 Day 1 | 6.681 [3.48 to 9.89] | -0.272 [-3.73 to 3.18]
  Cycle 51 Day 1 | 6.836 [3.51 to 10.16] | -0.363 [-3.95 to 3.23]
  Cycle 53 Day 1 | 6.990 [3.55 to 10.43] | -0.454 [-4.18 to 3.27]
  Cycle 55 Day 1 | 7.145 [3.58 to 10.71] | -0.544 [-4.40 to 3.31]
  Cycle 57 Day 1 | 7.300 [3.61 to 10.99] | -0.635 [-4.63 to 3.36]
  Cycle 59 Day 1 | 7.454 [3.64 to 11.26] | -0.726 [-4.86 to 3.41]
  Cycle 61 Day 1 | 7.609 [3.68 to 11.54] | -0.817 [-5.08 to 3.45]
  Cycle 63 Day 1 | 7.763 [3.71 to 11.82] | -0.907 [-5.31 to 3.50]
  Cycle 65 Day 1 | 7.918 [3.74 to 12.10] | -0.998 [-5.54 to 3.55]
Statistical Analysis 1: Comparison: Palbociclib + Letrozole vs Placebo + Letrozole; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.0078, Mixed effects model; Mean = 3.358, 95% CI 2-sided [0.88 to 5.83] — A positive change indicates improvement from baseline and a negative change indicates deterioration

22. Secondary Outcome: Model Estimated Mean Changes From Baseline in Functional Assessment of Cancer Therapy - Breast (FACT-B) Total Score
Description: The Functional Assessment of Cancer Therapy (FACT) is a modular approach to assess participant health related quality of life using a "core" set of questions (FACT-G) as well as a cancer site specific module. The FACT-G was a 27-item compilation of general questions divided into 4 domains: Physical Well Being, Social/Family Well Being, Emotional Well Being, and Functional Well Being. The FACT-B consists of the FACT-G (27 items) and a breast specific module: a 10-item instrument designed to assess participant concerns relating to breast cancer. For all questions, participants were asked to respond to a 5-level scale ranging from 0=Not at all to 4=Very much. FACT-B total score = FACT-G + Breast Cancer Subscale. As each of the items ranges from 0-4, the range of possible scores is 0-148, with 0 being the worst possible score and 148 the best. A positive change of the total score indicated improvement from baseline and a negative change indicated deterioration.
Time Frame: Baseline up to Cycle 65 Day 1
Population: This was a subset of intent-to-treat (ITT) population (participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or received a different drug from that to which they were randomized), who had both baseline and who completed >80% of the corresponding questions and had valid scores for the relevant subscales.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 166 | 171
Units on a scale
  Cycle 2 Day 1 | 1.618 [-0.15 to 3.39] | 1.021 [-0.74 to 2.78]
  Cycle 3 Day 1 | 1.441 [-0.32 to 3.20] | 0.850 [-0.90 to 2.60]
  Cycle 5 Day 1 | 1.087 [-0.69 to 2.86] | 0.510 [-1.25 to 2.27]
  Cycle 7 Day 1 | 0.732 [-1.07 to 2.53] | 0.169 [-1.62 to 1.96]
  Cycle 9 Day 1 | 0.378 [-1.48 to 2.23] | -0.171 [-2.02 to 1.68]
  Cycle 11 Day 1 | 0.024 [-1.90 to 1.95] | -0.512 [-2.44 to 1.41]
  Cycle 13 Day 1 | -0.331 [-2.34 to 1.68] | -0.852 [-2.88 to 1.17]
  Cycle 15 Day 1 | -0.685 [-2.80 to 1.43] | -1.193 [-3.33 to 0.95]
  Cycle 17 Day 1 | -1.039 [-3.27 to 1.19] | -1.534 [-3.80 to 0.74]
  Cycle 19 Day 1 | -1.393 [-3.75 to 0.96] | -1.874 [-4.29 to 0.54]
  Cycle 21 Day 1 | -1.748 [-4.24 to 0.75] | -2.215 [-4.78 to 0.35]
  Cycle 23 Day 1 | -2.102 [-4.74 to 0.54] | -2.555 [-5.28 to 0.17]
  Cycle 25 Day 1 | -2.456 [-5.24 to 0.33] | -2.896 [-5.79 to 0.00]
  Cycle 27 Day 1 | -2.810 [-5.76 to 0.13] | -3.326 [-6.31 to -0.16]
  Cycle 29 Day 1 | -3.165 [-6.27 to -0.06] | -3.577 [-6.83 to -0.33]
  Cycle 31 Day 1 | -3.519 [-6.79 to -0.25] | -3.918 [-7.35 to -0.48]
  Cycle 33 Day 1 | -3.873 [-7.31 to -0.43] | -4.258 [-7.88 to -0.64]
  Cycle 35 Day 1 | -4.227 [-7.84 to -0.62] | -4.599 [-8.41 to -0.79]
  Cycle 37 Day 1 | -4.582 [-8.37 to -0.80] | -4.939 [-8.95 to -0.93]
  Cycle 39 Day 1 | -4.936 [-8.90 to -0.97] | -5.280 [-9.48 to -1.08]
  Cycle 41 Day 1 | -5.290 [-9.43 to -1.15] | -5.620 [-10.02 to -1.22]
  Cycle 43 Day 1 | -5.644 [-9.97 to -1.32] | -5.961 [-10.56 to -1.36]
  Cycle 45 Day 1 | -5.999 [-10.50 to -1.50] | -6.301 [-11.10 to -1.50]
  Cycle 47 Day 1 | -6.353 [-11.04 to -1.67] | -6.642 [-11.64 to -1.64]
  Cycle 49 Day 1 | -6.707 [-11.58 to -1.84] | -6.983 [-12.18 to -1.78]
  Cycle 51 Day 1 | -7.061 [-12.12 to -2.00] | -7.323 [-12.73 to -1.92]
  Cycle 53 Day 1 | -7.416 [-12.66 to -2.17] | -7.664 [-13.27 to -2.05]
  Cycle 55 Day 1 | -7.770 [-13.20 to -2.34] | -8.004 [-13.82 to -2.19]
  Cycle 57 Day 1 | -8.124 [-13.74 to -2.51] | -8.345 [-14.37 to -2.32]
  Cycle 59 Day 1 | -8.478 [-14.29 to -2.67] | -8.685 [-14.91 to -2.46]
  Cycle 61 Day 1 | -8.833 [-14.83 to -2.84] | -9.026 [-15.46 to -2.59]
  Cycle 63 Day 1 | -9.187 [-15.37 to -3.00] | -9.367 [-16.01 to -2.72]
  Cycle 65 Day 1 | -9.541 [-15.92 to -3.16] | -9.707 [-16.56 to -2.86]
Statistical Analysis 1: Comparison: Palbociclib + Letrozole vs Placebo + Letrozole; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.7862, Mixed effects model; Mean = 0.476, 95% CI 2-sided [-2.97 to 3.92] — A positive change indicates improvement from baseline and a negative change indicates deterioration

23. Secondary Outcome: Median Baseline Percent (%) Positive Cells for Ki67
Description: Archived formalin-fixed paraffin embedded (FFPE) specimen from the original diagnostic tumor tissue was collected and sent to the sponsor-designated central laboratories for assessment of Ki67 associated with sensitivity and/or resistance to Palbociclib.
Time Frame: Baseline
Population: This was a subset of as-treated (AT) population (participants who received at least 1 dose of study medication, with treatment assignments designated according to actual study treatment received), who had both baseline and at least 1 follow-up values for Ki67.
Measure: Median (Full Range); unit: Percentage of Ki67 positive cells
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 146 | 156
Percentage of Ki67 positive cells | 30.0 [0 to 95] | 27.5 [0 to 95]

24. Secondary Outcome: Number of Participants With Detection in Estrogen Receptor (ER)
Description: Archived formalin-fixed paraffin embedded (FFPE) specimen from the original diagnostic tumor tissue was collected and sent to the sponsor-designated central laboratories for assessment of ER associated with sensitivity and/or resistance to Palbociclib.
Time Frame: Baseline
Population: This was a subset of as-treated (AT) population (participants who received at least 1 dose of study medication, with treatment assignments designated according to actual study treatment received), who had both baseline and at least 1 follow-up values for ER.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 168 | 171
Participants
  Positive | 152 | 162
  Negative | 2 | 1
  Unknown | 14 | 8

ADVERSE EVENTS:
Time Frame: 65 months
Description: Participants were only counted once per treatment for each category
Arm/Group | Palbociclib + Letrozole | Placebo + Letrozole
All-Cause Mortality (participants affected / at risk) | 79/168 | 86/171
Serious Adverse Events (participants affected / at risk) | 26/168 | 16/171
Other Adverse Events (participants affected / at risk) | 168/168 | 142/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib + Letrozole (N=168) | Placebo + Letrozole (N=171)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Ear disorder (Ear and labyrinth disorders) | 0 | 1
Thyroid mass (Endocrine disorders) | 0 | 1
Clinical death (General disorders) | 1 | 0
Disease progression (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Liver injury (Hepatobiliary disorders) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Platelet count decreased (Investigations) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ovarian cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib + Letrozole (N=168) | Placebo + Letrozole (N=171)
Anaemia (Blood and lymphatic system disorders) | 65 | 13
Leukopenia (Blood and lymphatic system disorders) | 48 | 8
Neutropenia (Blood and lymphatic system disorders) | 74 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 23 | 0
Cataract (Eye disorders) | 12 | 10
Lenticular opacities (Eye disorders) | 9 | 7
Constipation (Gastrointestinal disorders) | 6 | 10
Diarrhoea (Gastrointestinal disorders) | 18 | 14
Mouth ulceration (Gastrointestinal disorders) | 13 | 0
Nausea (Gastrointestinal disorders) | 16 | 15
Toothache (Gastrointestinal disorders) | 10 | 3
Fatigue (General disorders) | 17 | 14
Influenza like illness (General disorders) | 13 | 8
Oedema peripheral (General disorders) | 9 | 6
Pain (General disorders) | 10 | 13
Pyrexia (General disorders) | 24 | 10
Nasopharyngitis (Infections and infestations) | 13 | 10
Upper respiratory tract infection (Infections and infestations) | 19 | 20
Alanine aminotransferase increased (Investigations) | 56 | 56
Aspartate aminotransferase increased (Investigations) | 58 | 48
Bilirubin conjugated increased (Investigations) | 11 | 7
Blood alkaline phosphatase increased (Investigations) | 9 | 14
Blood bilirubin increased (Investigations) | 11 | 13
Blood creatinine increased (Investigations) | 10 | 2
Blood lactate dehydrogenase increased (Investigations) | 11 | 8
Electrocardiogram QT prolonged (Investigations) | 25 | 14
Gamma-glutamyltransferase increased (Investigations) | 17 | 12
Haemoglobin decreased (Investigations) | 19 | 3
Low density lipoprotein increased (Investigations) | 8 | 9
Neutrophil count decreased (Investigations) | 110 | 19
Platelet count decreased (Investigations) | 70 | 7
Red blood cell count decreased (Investigations) | 10 | 2
Weight increased (Investigations) | 18 | 12
White blood cell count decreased (Investigations) | 106 | 15
Hyperglycaemia (Metabolism and nutrition disorders) | 16 | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 12 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 18 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 12
Dizziness (Nervous system disorders) | 17 | 11
Headache (Nervous system disorders) | 13 | 7
Insomnia (Psychiatric disorders) | 10 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 22
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 20 | 11
Rash (Skin and subcutaneous tissue disorders) | 11 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2014-07-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT02297438/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT02297438/SAP_001.pdf